CLINICAL TRIAL: NCT03219840
Title: Effects of Cetylpyridium Chloride (CPC) Based Chewing Gum Plus Tooth Brushing on Plaque Formation and Gingivitis: a Randomized, Double-Blind, Crossover, Placebo-controlled Clinical Trial
Brief Title: Cetylpyridium Chloride (CPC) Based Chewing Gum and Gingivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: CONFADENT Oral Technology, Kiss Industries LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSC-DB-17-0313
Record Dates: First submitted 2017-07-13; First posted 2017-07-18 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Gingivitis; Plaque, Dental; Periodontal Diseases
Keywords: Cetylpyridium Chloride (CPC); Chewing Gum
MeSH Terms: conditions — Gingivitis; Dental Plaque; Periodontal Diseases | interventions — Cetylpyridinium; cytidylyl-(3'-5')-cytidine

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-blind, Crossover, Placebo-controlled Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPC + Xylitol chewing gum, then Xylitol only chewing gum (Experimental): Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum and then Xylitol only chewing gum All subjects will be instructed to chew four times a day, for at least 60 seconds, after which they expectorated. Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum will be used for the first 21 days, then there will be a washout period of 21 days, and finally Xylitol only chewing gum will be used for the last 21 days.
  Interventions: Drug: Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum; Drug: Xylitol only chewing gum
- Xylitol only chewing gum, then CPC + Xylitol chewing gum (Experimental): Xylitol only chewing gum and then Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum All subjects will be instructed to chew four times a day, for at least 60 seconds, after which they expectorated. Xylitol only chewing gum will be used for the first 21 days, then there will be a washout period of 21 days, and finally Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum will be used for the last 21 days.
  Interventions: Drug: Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum; Drug: Xylitol only chewing gum

INTERVENTIONS:
Drug: Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum — All subjects will be instructed to chew four times a day, for at least 60 seconds, after which they expectorated.
Drug: Xylitol only chewing gum — All subjects will be instructed to chew four times a day, for at least 60 seconds, after which they expectorated.

SUMMARY:
This placebo-controlled, double-blinded, randomized crossover study evaluates the plaque and gingivitis reducing capacity of Cetylpyridium Chloride (CPC) chewing gum, with mechanical oral hygiene. The study will enroll 73 students, faculty, and staff from the UTHealth School of Dentistry. Half of the eligible participants will be randomly assigned to get the CPC gum in the first treatment period (21 days), a wash-out period of 21 days, and then a placebo gum in the second treatment period (21 days). The other half will be assigned to follow the same schedule but with the treatment reversed. A statistician will perform the randomization. Primary outcomes are assessed by validated tools, such as the Plaque Index (PI), Gingival Index (GI), and percent of bleeding sites on probe (BOP).

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 and older
* Be capable of giving informed consent themselves and are able and willing to participate in the study
* Patients willing to forgo any optional dental procedures during the study period, such as dental prophylaxis or teeth whitening
* Patients that regularly brush their teeth twice a day

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients taking long-term anti-microbial or anti-inflammatory drugs
* Patients unable or unwilling to provide informed consent
* Self-reported use of tobacco products
* Gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque or calculus, or soft or hard tissue tumor of the oral cavity
* Less than 26 teeth in the mouth
* Orthodontic appliances or removable partial dentures that will compromise the ability of the potential subject to participate in the study
* Periodontitis as indicated periodontal pockets greater than 5 millimeters on more than one site
* Inability to comply with assigned treatment regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2018-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Lakschevitz, DDS, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was enrolled but then was lost to follow up before randomization.
Groups:
- CPC + Xylitol Chewing Gum, Then Xylitol Only Chewing Gum: Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum, and then Xylitol only chewing gum All subjects will be instructed to chew four times a day, for at least 60 seconds, after which they expectorated. Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum will be used for the first 21 days, then there will be a washout period of 21 days, and finally Xylitol only chewing gum will be used for the last 21 days.
- Xylitol Only Chewing Gum, Then CPC + Xylitol Chewing Gum: Xylitol only chewing gum, and then Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum All subjects will be instructed to chew four times a day, for at least 60 seconds, after which they expectorated. All subjects will be instructed to chew four times a day, for at least 60 seconds, after which they expectorated. Xylitol only chewing gum will be used for the first 21 days, then there will be a washout period of 21 days, and finally Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum will be used for the last 21 days.
Period: Overall Study
Arm/Group | CPC + Xylitol Chewing Gum, Then Xylitol Only Chewing Gum | Xylitol Only Chewing Gum, Then CPC + Xylitol Chewing Gum
Started | 38 | 31
Day 1 Visit for 1st Period | 37 | 31
1st Intervention Period of 21 Days | 34 | 31
Day 22 Visit for 1st Period | 34 | 31
Washout Period of 21 Days | 34 | 31
Day 1 Visit for 2nd Period | 34 | 31
2nd Intervention Period of 21 Days | 34 | 31
Day 22 Visit for 2nd Period | 34 | 31
Completed | 34 | 31
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum will be used during one period of 21 days and Xylitol only chewing gum will be used during another period of 21 days, with the two periods divided by a washout period of 21 days. All subjects will be instructed to chew four times a day, for at least 60 seconds, after which they expectorated.
Arm/Group | All Participants
Number analyzed (Participants) | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 69
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Degree of Plaque as Assessed by the Turesky Modification of the Quigley-Hein Plaque Index
Description: Plaque will be assessed using the Turesky Modification of the Quigley-Hein Plaque Index, where a score of 0 to 5 will be assigned to each facial and lingual non-restored surface of all teeth that are present with the exception of third molars at baseline and week 3 of the study, as follows. For each participant, an average of the scores for all teeth is calculated.
  0 No plaque
  1. Separate flecks of plaque at the cervical margin of the tooth
  2. A thin continuous band of plaque (up to one mm) at the cervical margin of the tooth
  3. A band of plaque wider than one mm but covering less than one-third of the crown of the tooth
  4. Plaque covering at least one-third but less than two-thirds of the crown of the tooth
  5. Plaque covering two-thirds or more of the crown of the tooth
Time Frame: day 1
Population: For each arm, 2 participants were lost to follow up. Also, for each arm, 2 other participants did not follow the protocol, and their data were not analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cetylpyridinium Chloride (CPC) 0.09% + Xylitol Chewing Gum: Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum will be used for a period of 21 days. All subjects will be instructed to chew four times a day, for at least 60 seconds, after which they expectorated.
- Xylitol Only Chewing Gum: Xylitol only chewing gum will be used for a period of 21 days. All subjects will be instructed to chew four times a day, for at least 60 seconds, after which they expectorated.
Arm/Group | Cetylpyridinium Chloride (CPC) 0.09% + Xylitol Chewing Gum | Xylitol Only Chewing Gum
Number analyzed (Participants) | 65 | 65
score on a scale | 0.41 (0.28) | 0.43 (0.28)

2. Primary Outcome: Degree of Plaque as Assessed by the Turesky Modification of the Quigley-Hein Plaque Index
Description: as for outcome 1
Time Frame: day 22
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cetylpyridinium Chloride (CPC) 0.09% + Xylitol Chewing Gum | Xylitol Only Chewing Gum
Number analyzed (Participants) | 65 | 65
score on a scale | 0.36 (0.26) | 0.35 (0.28)

3. Primary Outcome: Degree of Gingivitis as Assessed by the Gingival Index (GI)
Description: Gingivitis will be assessed using the Gingival Index (GI), where a score of 0 to 3 will be assigned to six teeth, representing six segments of jaws, at baseline and week 3 of the study according to the following criteria. For each participant, an average of the scores for all 6 teeth is calculated.
  0 Absence of inflammation.
  1. Mild inflammation - slight change in color and little change in texture.
  2. Moderate inflammation - moderate glazing, redness, edema, and hypertrophy. Bleeding on pressure.
  3. Severe inflammation - marked redness and hypertrophy. Tendency to spontaneous bleeding. Ulceration.
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cetylpyridinium Chloride (CPC) 0.09% + Xylitol Chewing Gum | Xylitol Only Chewing Gum
Number analyzed (Participants) | 65 | 65
score on a scale | 0.16 (0.41) | 0.19 (0.40)

4. Primary Outcome: Degree of Gingivitis as Assessed by the Gingival Index (GI)
Description: as for outcome 3
Time Frame: day 22
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cetylpyridinium Chloride (CPC) 0.09% + Xylitol Chewing Gum | Xylitol Only Chewing Gum
Number analyzed (Participants) | 65 | 65
score on a scale | 0.21 (0.64) | 0.15 (0.34)

5. Primary Outcome: Degree of Gingival Bleeding as Assessed by the Bleeding on Probing (BOP) Index
Description: Bleeding on probing (BOP) as described in Ainamo & Bay 1975 will be assessed, where each of 4 gingival areas (disto-buccal, midbuccal, mid-lingual, and mesio-lingual) around each tooth will be light probed and scored from 0 to 2 as follows. For each participant, an average of the scores for the 4 gingival areas is calculated.
  0 Absence of bleeding after 30 seconds
  1. Bleeding after 30 seconds
  2. Immediate bleeding
Time Frame: day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cetylpyridinium Chloride (CPC) 0.09% + Xylitol Chewing Gum | Xylitol Only Chewing Gum
Number analyzed (Participants) | 65 | 65
score on a scale | 0.09 (0.06) | 0.11 (0.09)

6. Primary Outcome: Degree of Gingival Bleeding as Assessed by the Bleeding on Probing (BOP) Index
Description: Bleeding on probing (BOP) as described in Ainamo & Bay 1975 will be assessed, where each of 4 gingival areas (disto-buccal, midbuccal, mid-lingual, and mesio-lingual) around each tooth will be light probed and scored from 0 to 2 as follows. For each participant, an average of the scores for all teeth is calculated, an average of the scores for the 4 gingival areas is calculated.
  0 Absence of bleeding after 30 seconds
  1. Bleeding after 30 seconds
  2. Immediate bleeding
Time Frame: day 22
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cetylpyridinium Chloride (CPC) 0.09% + Xylitol Chewing Gum | Xylitol Only Chewing Gum
Number analyzed (Participants) | 65 | 65
score on a scale | 0.08 (0.08) | 0.09 (0.09)

7. Secondary Outcome: Discoloration of Teeth as Assessed by the Vita Scale
Description: Objective observation of Discoloration of teeth will be recorded using a Vita scale. The color of the participant's teeth is matched to the colors on the scale. The colors in the scale are A1, A2, A3, A3.5, A4, B1, B2, B3, B4, C1, C2, C3, C4, D2, D3, and D4--the letter portion of the scale indicates a tooth color of reddish-brownish (A), reddish-yellowish (B), greyish (C), or reddish-grey (D), and the number portion of the scale indicates degree of discoloration, with 1 indicating least discoloration and 4 indicating the most discoloration.
Time Frame: day 1
Population: For each arm, data were not collected for 7 participants (2 of which were lost to follow up), and 2 other participants did not follow the protocol and their data were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetylpyridinium Chloride (CPC) 0.09% + Xylitol Chewing Gum | Xylitol Only Chewing Gum
Number analyzed (Participants) | 60 | 60
Participants
  A1 | 28 | 30
  A2 | 21 | 19
  A3 | 4 | 1
  A3.5 | 0 | 3
  A4 | 0 | 0
  B1 | 6 | 6
  B2 | 1 | 0
  B3 | 0 | 0
  B4 | 0 | 0
  C1 | 0 | 1
  C2 | 0 | 0
  C3 | 0 | 0
  C4 | 0 | 0
  D2 | 0 | 0
  D3 | 0 | 0
  D4 | 0 | 0

8. Secondary Outcome: Discoloration of Teeth as Assessed by the Vita Scale
Description: as for outcome 7
Time Frame: day 22
Population: Data were not collected for 5 in the Cetylpyridinium Chloride (CPC) 0.09% + Xylitol chewing gum arm (2 of which were lost to follow up). Data also were not collected for 3 in the Xylitol only chewing gum arm (2 of which were lost to follow up). For each arm, 2 other participants did not follow the protocol, and their data were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetylpyridinium Chloride (CPC) 0.09% + Xylitol Chewing Gum | Xylitol Only Chewing Gum
Number analyzed (Participants) | 62 | 64
Participants
  A1 | 25 | 27
  A2 | 24 | 22
  A3 | 3 | 2
  A3.5 | 1 | 0
  A4 | 0 | 0
  B1 | 8 | 10
  B2 | 0 | 1
  B3 | 0 | 0
  B4 | 0 | 0
  C1 | 0 | 0
  C2 | 0 | 1
  C3 | 0 | 0
  C4 | 0 | 0
  D2 | 0 | 1
  D3 | 1 | 0
  D4 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through the day 22 visit of second intervention period
Description: For each arm, 2 participants were lost to follow up, and 2 participants were removed from the study for not following the protocol.
Arm/Group | Cetylpyridinium Chloride (CPC) 0.09% + Xylitol Chewing Gum | Xylitol Only Chewing Gum
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT03219840/Prot_SAP_000.pdf